CLINICAL TRIAL: NCT06705348
Title: Role of Synaptic Density in Mediating the Relation Between Social Disconnection and Late-life Suicide Risk
Brief Title: Social Disconnection Study
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Irina Esterlis, Professor of Psychiatry, Yale University
Other Study IDs: 2000033973
Record Dates: First submitted 2024-11-12; First posted 2024-11-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Social Disconnection
Keywords: loneliness; social disconnection; isolation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood may be collected for genetic testing of APOE (a gene associated with Alzheimer's disease) and for DNA testing of polymorphisms in genes of interest to mental health.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Transdiagnostic: Participants will be a transdiagnostic sample of older individuals (age 55+ years) with stress disorders without psychosis including individuals with MDD, bipolar disorder, post-traumatic stress disorder (PTSD), dysthymia, and non-psychiatric individuals.

SUMMARY:
The purpose of this research study is to examine the effect of social connectedness on the brain. Study procedures include one Magnetic Resonance Imaging (MRI) or functional Magnetic Resonance Imaging (fMRI) scan, one Positron Emission Tomography (PET) scan, one Magnetic Resonance Spectroscopy (MRS) scan, an electroencephalogram (EEG), and in-person and phone call follow-ups.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effect of social connectedness (social isolation and loneliness) on synaptic density in the brain using PET scans. Participants will have a screening appointment to determine eligibility. Participants will participate in the following study procedures:

MRI or fMRI scan: the purpose of the MR scan is to help us identify the different regions of the brain on the PET scans. Participants may be asked to do some cognitive and behavioral tasks during parts of the MR scan.

PET scan: an arterial catheter and one or two IV catheters will be placed (one for radiotracer injection and one to take blood samples). The radiotracer, [18F]SDM-8 will be used. A radiotracer is a minimal amount of a drug that is labeled with a very small amount of a radioactive substance that binds to receptors in the brain and can be detected by a special camera in the PET scanner.

Electroencephalography (EEG): EEG is a procedure that allows measurement of physiological brain responses. Sensors placed on and around the head record small electrical currents produced by the brain.

Follow-up phone calls and appointments: participants will have follow-up phone calls every 3 months for 9 months following scan visits, and an in-person follow-up appointment 1 year after scans to assess mood and cognition, as well as document any changes. Follow-up assessments may continue for up to 5 years after the year one follow-up appointment.

Some subjects may be asked to return after the 1 year follow-up period to repeat study procedures to examine changes over time.

ELIGIBILITY:
Inclusion Criteria:

* able to give written informed consent
* age 55+
* English speaking

Exclusion Criteria:

* contraindication to MRI scanning including claustrophobia, high girth, moderate to significant white matter atrophy, and presence of ferromagnetic material in the body, including orthodontic braces or other non MR-compatible foreign bodies. All participants will be screened for metal objects by the same methods used for routine clinical MRI scanning
* for women: pregnancy or breastfeeding
* serious medical or neurological illness that in the opinion of the PI would interfere with the scientific goals of the study or participant safety
* pervasive developmental disorders (PDD) or primary psychotic disorders
* meet DSM-5 criteria for current severe substance use disorder (except marijuana or nicotine)
* head injury that led to significant long term decline in cognitive abilities as seen by decline in grades or work performance
* current psychosis, active significant suicidal (score of 6 on MADRS suicide item) or homicidal ideation
* lifetime history of neurologic abnormality including seizure disorder, cerebrovascular, or neoplastic lesion, neurodegenerative disorder, or significant head trauma resulting in post-traumatic amnesia >24 hours
* full scale IQ lower than 70
* contraindications to PET (e.g. poor venous access for placement of venous lines)
* history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year
* history of a bleeding disorder or currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto) *for subjects obtaining arterial line.
* blood donation within 8 weeks of the start of the study
* REM sleep disorder
* brain injury (TBI, seizure/epilepsy, stroke, TIA) in lifetime (self-report and medical chart review)
* electroconvulsive or ketamine therapy, or similar therapies that have rapid effects on brain neurochemistry within the past 6 months
* high risk for stroke (above first quartile on Framingham Stroke Risk Profile)
* current cancer

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Transdiagnostic sample of older individuals (age 55+ years) with stress disorders without psychosis including individuals with MDD, bipolar disorder, post-traumatic stress disorder (PTSD), dysthymia, and non-psychiatric individuals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Social disconnection | enrollment to end of study participation (approximately 1 year)
  Social disconnection composite measure determined by the following:
  Item #3 - Hamilton Depression Rating Scale (social withdrawal; range = 0-4) Item #12 - Beck Depression Inventory-II (loss of interest in people; range = 0-3) Item #14 - Center for Epidemiologic Studies Depression Scale (feelings of loneliness; range = 0-3) Item #2 - Snaith-Hamilton Pleasure Scale (enjoyment being with family or close friends; range = 0-1) Item #7 - Snaith-Hamilton Pleasure Scale (enjoyment seeing other people's smiling faces; range = 0-1) Item #17 - Profile of Mood States (loneliness; range = 0-4)
  Higher composite score = greater severity of social disconnection.
SV2A density | enrollment to end of study participation (approximately 1 year)
  SV2A density as measured using [18F]SDM8 PET imaging.

SECONDARY OUTCOMES:
Composite measure of suicide risk | enrollment to end of study participation (approximately 1 year)
  Suicide risk will be operationalized as a composite score of death ideation, depressive symptoms, loss of personal and self-worth, executive control, and perceived meaning in life based on the following:
  Geriatric Suicide Ideation Scale (GSIS) suicide ideation subscale score (range 10-50, higher score indicates greater active suicidal ideation).
  GSIS death ideation subscale score (range 5-25, higher score indicates greater death ideation) Montgomery Asberg Depression Rating Scale (MADRS) total score (range 0-60, higher score indicates greater severity of depression) GSIS loss of personal and social worth subscale score (range 7-35, higher score indicates greater feeling of loss of personal and social worth) Cogstate Go/No-Go task score GSIS perceived meaning in life subscale score (range 8-40, higher score indicates lower perceived meaning in life)
Sex | enrollment to end of study participation (approximately 1 year)
Composite measure of suicide risk over time | 12-month study period (from scanning to year 1 follow-up)
  identification of predominant trajectories of suicide risk measures (see 'composite measure of suicide risk' outcome measure) over 5 time points spanning the 12-month study period (0, 3, 6, 9, and 12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Irina Esterlis, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Translational Brain Imaging Program, New Haven, Connecticut, United States